CLINICAL TRIAL: NCT03397823
Title: The Characterisation of Therapeutic Radiation-induced Caries; the Histopathological, Ultrastructural and Microbial Changes Affecting Its Prevention and Treatment.
Brief Title: The Characterisation of RT Caries.
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Other Study IDs: Radiotherapy caries
Record Dates: First submitted 2017-12-14; First posted 2018-01-12 (Actual); Last update posted 2021-09-13 (Actual); Status verified 2018-12

CONDITIONS: Head and Neck Cancer; Radiotherapy Side Effect
MeSH Terms: conditions — Head and Neck Neoplasms; Radiation Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- head and neck cancer pre RT: head and neck cancer patients before and after RT
- head and neck cancer treated: head and neck cancer patients treated with radiotherapy
- control group: age gender matched subjects

SUMMARY:
Overcoming limitations of previous studies, the following research project will assess the most significant acute and long-term complications of RT that affect HNC patients: oral mucositis, dry mouth feeling, taste alteration and carious lesion incidence, all of which negatively affect cancer treatment outcomes and the quality of life of cancer survivors. This project was developed with an aim to study any possible correlations / links between the oral sequelae of RT and the negative clinical outcomes listed, in order to help the development of clinical management protocols for HNC patients to mitigate the effect on care and patient comfort and its delivery in healthcare systems.

The project comprises of a longitudinal cohort study of HNC patients correlating biodata of biochemical salivary parameters, clinical outcomes and oral health status over a period up to 12 months post-RT, focusing on baseline pre-IMRT (T0), 6 months post-IMRT (T1) and up to 12 months post-IMRT treatments (T2). The ultimate goal is to identify possible predictive markers in the saliva at T0 to assist with evaluation of oral mucositis severity in individual HNC patients prior to start of treatment so that treatment can be adapted for such high-risk patients individually, to either prevent or minimise the severity of this consequence of RT.

DETAILED DESCRIPTION:
1. Introduction

   Head and neck cancer is the sixth most common cancer in the world representing 4-5% of all malignancies . Head and neck cancer (includes oral, nasal cavity, salivary glands, paranasal sinus, pharynx, and larynx) is one of the top 10 most diagnosed cancers in the UK . According to Cancer Research UK, there were 7591 newly diagnosed with oral cancer in 2013 in the country, representing the 14th most common cancer in the UK.

   Radiotherapy (RT) is the first choice treatment for the majority head and neck cancer patients, which is a localized treatment to control the tumour . More than 50% of head and neck cancer patients receive RT delivered in fractions of 2 Grays (Gy) daily during 5 days per week until the end of their therapy dosage (mean cumulative dose 55-77 Gy). RT stimulates cellular changes that destroy the tumor cells, but may affect dramatically the healthy oral tissues altering the homeostasis of this complex environment. RT is the cause of a wide range of adverse oral tissue reactions such as permanent damage of the major and minor salivary glands (hyposalivation, xerostomia), modification of connective and vascular tissues and a reduction the healing capacity especially in mucosal and mineralised tissues (mucositis, caries lesion, osteoradionecrosis). In order to try to diminish the adverse side effects of the RT three-dimensional (3D) computed tomography (CT) planned radiotherapy known as intensity-modulated radiotherapy (IMRT) has been developed .

   There are acute (mucositis) and late-onset adverse effects/sequelae that RT induces in healthy oral tissues . Radiation-induced dental caries is the most common late effect, but its origin and nature is not clear. RT related caries have a rapid onset as a result of a combination of factors such as shift in oral microbial community composition favouring acidophilic bacteria, hypo-salivation, poor oral hygiene and dietary alterations . The patients often have little/no pain, even in the most severe cases. Histological features show that the onset and development of caries is similar to non RT-related ones but the sites affected are different. Indeed RT-related caries is more frequent on the cervico-labial surface/ incisal edge of canines and incisors while non RT-related ones are more frequent in the interproximal/ occlusal areas of the posterior teeth (molar and premolars).

   Also, caries associated with RT has a rapid circumferential progression which may lead to tooth fracture. It is characterized by a localized lesion to the incisal or occlusal surfaces which diffuse and progress in relation to irregular and generalized erosion of the incisal edge of the tooth. In addition, mechanical changes (increased elastic modulus and stiffness) within the tooth structure increase the wear of the incisal and occlusal areas and could lead to complete fracture of the tooth.

   Tooth destruction is one of the most severe consequences of RT and it may produce complete edentulousness in 3 - 5 years. The dental management of RT patients is challenging. It is necessary to gather a multidisciplinary team (restorative dentists, periodontology, endodontic, dental hygienist, radiation oncologists, medical oncologists, and oral surgeons) to maintain oral health and improve quality of life (QoL). Almost 50% of cancer survivors reported depression, worry or tension related to oral dryness symptoms. Hence, RT sequelae detrimentally affect the quality of life of head and neck cancer patients.

   Overall, it is necessary the quantitative analysis of chemical matrix components, proteins and microbial changes that occur in patients' teeth/oral cavity, who have undergone RT, in order to determine the aetiology and pathophysiology of the two prevalent side effects (caries/mucositis) to correlate with preventive measurement and appropriate treatment care for this population. Finally, it is necessary to perform a complete oral assessment using a validated index in order to create a baseline record before the treatment and a validated measured to compare after the RT and with healthy individuals.
2. Aim The aim of this project is to perform a well-controlled and integrated longitudinal study of HNC patients correlating biodata of biochemical parameters, clinical parameters and oral health status, to overcoming the limitations of previous studies, that examined the different side effects of radiotherapy of HNC patients (reduced number, retrospective, observational, short term follow up, lack of detailed clinical assessment, focused into treatment of side effects).

   The first objective of this study will be to perform quantitative analysis of oral/ dental status of HNC patients pre and post IMRT and analyse the possible associations between the clinical outcomes.

   Followed by assessing salivary gland function of HNC patients pre and post IMRT by analysing protein concentration and secretion rate and investigate the possible associations between these proteins and clinical outcomes.

   Next objective is to determine the possible association between selected proteins concentration and secretion rate and oral mucositis outcomes after IMRT, and therefore, the final objective is to evaluate whether protein concentration or secretion rate of saliva is a reliable predictor of mucositis presence and severity.

   Null Hypothesis There will be no correlation between salivary biochemical composition and oral side effects of radiotherapy in the HNC patients before and after radiotherapy
3. Materials and Methods. Ethics application to Health Research Authority (IRAS Project ID:199100). All the samples of the study would be obtained from the Special Care dental Unit at KCL Dental Institute, Guy's Hospital and from the Dental Clinic at KCL Dental Institute.

The samples will include saliva, biofilm, mucosal swabs, carious dentine and/or teeth. The samples collection will add approximately 10 to 20 min to the conventional treatment time. All the samples will be collected at 3-time points before and after IMRT from the head and neck cancer up to 12 months follow up.

Patients over the age of 18 in order to analyse permanent dentition and the age range for cancer patients are over 18 years old, both gender,at any stage of disease, except where distant metastases.

Subjects withouth Head and neck cancer age and gender matched. Following these inclusion criteria the next patients are excluded younger than 18 (non-permanent dentition), unable to give the consent patients who have been administered antibiotics in the previous 3 months because the oral microbiota could be altered , patients with systemic disease (such as Sjogren syndrome), subjects with non-controlled systemic diseases, that can affect the salivary flow and host defence mechanism.

Sample size Calculation Statement Statistical advice was obtained prior to start this study in order to determine the sample size required by a suitable power calculation. The power calculation was based on comparing the mean protein levels in head and neck cancer patients before and after IMRT. A study with 80% power at 5% level of significance (Chaudhury et al., 2015) will be able to detect the true difference in all parameters before and after cancer treatment with an effect size of 0.5 (high according to Cohen 1988) using two tailed test would require a total sample of 35 patients

Proposed statistical analysis:

Descriptive statistics will be used to summarize the sample characteristics and other clinical factors.

All analysis will be carried out using STATA 15.1 (College Station, Texas USA, www.stata.com), GraphPad Prism 8 software (La Jolla California USA, www.graphpad.com) and Microsoft Excel 2018, after checking for normality. Normality of the data will be tested for all the parametric analyses using histogram and box plots. Results expresses as a mean ± SEM relative to the variables and 'n' represents the number of subjects, p <0.05 value was considered statistically significant.

Sample Collection

The following samples will be collected:

* unstimulated whole mouth saliva (UWMS), saline solution rinse
* plaque biofilm
* mucosal swabs collecting residual saliva from the inner cheek
* excavated carious dentine tissue and/or extracted carious teeth. Sample collection will add 15 min to the conventional treatment time. Samples will be collected during the day, routinely between the hours 1:30pm to 3:30pm in the dental clinic in an attempt to avoid diurnal variations.

Unstimulated Whole Mouth Saliva Sample Collection (UWMS)

UWMS samples will be obtained by passive drooling into a pre -weighed 50 mL sterile conical polypropylene tube (Falcon; BD Biosciences, San Jose, CA, USA) for 10 minutes. All participants will avoid food and drink for at least 60 min prior to sample collection. The samples wll be kept on ice at 4°C, After collection, the tubes will be re-weighed and the net saliva volume calculated. Saliva samples will be labelled and stored in - 80 °C freezers for further analysis. Saliva flow rate will be calculated.

Clinical Oral Assessment Dry Mouth and Taste Report answering a question from a validated questionaire by Fox et al (Fox et al., 1987) and a question extracted from the Late Effects of Normal Tissue/Somatic Objective Management Analytic (LENT/SOMA) scoring system.

Oral Mucositis Grading using The World Health Organization (WHO) Oral Toxicity Scale Dental Assessment of carious lesions present from clinically visible change of colour to dark brown on any surface to open lesions in the oral cavity. Number of teeth / decayed, missed or filled (DMFT) will be included in the clinical assessment.

Sample Analysis

UWMS saliva samples Samples will be analysed for total protein content using the Bicinchoninic Acid Assay (BCA), targeted protein concentration by Enzyme-Linked Immunosorbent Assay (ELISA), Periodic Acid Schiff (PAS) staining, Coomassie Brilliant blue and α-amylase activity by the standard kinetic enzyme assay (Salimetrics).

Prior to biochemical analysis UWMS samples will be centrifuged at 10000 RPM for 5 mins at 4°C. The supernatant will be separated to be used to analyse protein content and the pellet was preserved to perform DNA extraction.

Protein Analysis (Concentration and Secretion Rate) Mucin 5B mucin 7, IgA, α-amylase, albumin carbonic anhydrase VI, acidic proline rich protein and statherin were selected due to their relationship to host defence, antimicrobial, bacterial adherence, colonization, mucosal pellicle, enamel pellicle, viscoelastic, rheological properties, lubrication, and remineralization.

Total protein secretion rate will be calculated by multiplication of the salivary flow rate and protein concentration in ug / min (Carpenter et al., 2000).

Mucin 5B and 7 will be quantified by PAS,α-amylase by a kinetic assay,IgA, albumin, cystatin S, proline rich protein and statherin concentration in UWMS will be determined using ELISA.

ELIGIBILITY:
Inclusion Criteria:

Head and Neck Cancer Patients Male or female Over the age of 18. Received radiation treatment for Head and Neck cancer

Exclusion Criteria:

Subjects younger than 18. Patients unable to give consent. Patients with non-controlled systemic disease Distant metastases Patients who have been administered antibiotics in the previous 3 months Patients with Sjogren syndrome. Patients with Rheumatoid arthritis Neurological disorders (Parkinson's disease) Dehydration Sialoadenitis Sialolithiasis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Head and neck cancer patients treated with radiotherapy
Sampling Method: Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2017-02-15 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
Effects of IMRT on saliva composition and potential associations with oral side effects | october 2019
  integrated longitudinal study of HNC patients correlating biodata of biochemical parameters, clinical parameters and oral health status

SECONDARY OUTCOMES:
IMRT effects on oral cavity | 2019
  to develop a quantitative analysis of oral/ dental status of HNC patients pre and post IMRT and analyse the possible associations between the clinical outcomes.
IMRT effects on biochemical composition of saliva | 2019
  to asses salivary gland function of HNC patients pre and post IMRT by analysing protein concentration and secretion rate and investigate the possible associations between these proteins and clinical outcomes
Association between selected salivary proteins and oral mucositis outcomes after IMRT | 2019
  To correlate biodata of biochemical salivary parameters, clinical outcomes and oral health status over a period up to 12 months post-RT in order to to identify possible predictive markers in the saliva for mucositis severity

CONTACTS AND LOCATIONS:
Overall Officials: avijit banerjee, professor, Principal Investigator — King's College London
Locations (1):
- kings college london, Guy's Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
the participants are allocated with a number its not possible to identify them